CLINICAL TRIAL: NCT04454515
Title: The Effect of Intraoperative Dexmedetomidine on Postoperative Morphine Requirements and Oral Intake After Breast Cancer Surgery
Brief Title: The Effect of Intraoperative Dexmedetomidine on Postoperative Morphine Requirements After Breast Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202004120MINB
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-01

CONDITIONS: Morphine Consumption
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: one group is going to receive precedex and another is placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexmedetomidine (Experimental): patient recieving dexmedetomidine
  Interventions: Drug: Dexmedetomidine
- placebo (Placebo Comparator): patients receiving placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine is an α2 receptor agonist with sedative and analgesic properties. In previous reports, dexmedetomidine improves smoothness of postoperative recovery and reduces intraoperatory imflammatory responses. As patients receiving breast surgeries are especially vulnerable to postoperative nausea/ vomiting, the dosage of narcotics and associated complications were concerned for not only comfortness but also postoperative oral intake and discharge.
  Arms: dexmedetomidine
Drug: placebo — normal saline infusion
  Arms: placebo

SUMMARY:
Dexmedetomidine is an α2 receptor agonist with sedative and analgesic properties. In previous reports, dexmedetomidine improves smoothness of postoperative recovery and reduces intraoperatory imflammatory responses. As patients receiving breast surgeries are especially vulnerable to postoperative nausea/ vomiting, the dosage of narcotics and associated complications were concerned for not only comfortness but also postoperative oral intake and discharge. The invetigators aimed to compare the effects of dexmedetomidine infusion versus placebo on postoperative narcotics requirement, complications, and oral intake.

DETAILED DESCRIPTION:
Dexmedetomidine is an α2 receptor agonist with sedative and analgesic properties. In previous reports, dexmedetomidine improves smoothness of postoperative recovery and reduces intraoperatory imflammatory responses. As patients receiving breast surgeries are especially vulnerable to postoperative nausea/ vomiting, the dosage of narcotics and associated complications were concerned for not only comfortness but also postoperative oral intake and discharge.

The invetigators aimed to compare the effects of dexmedetomidine infusion versus placebo on postoperative narcotics requirement, complications, and oral intake.

The participantss under general anesthesia and aged from 30 to 65 years old will be enrolled. All subjects were randomized into the dexmedetomidine or placebo group. They received placebo (group P, n = 30) or dexmedetomidine (loading dose of 1 μg kg-1 followed by 0.5 μg kg-1 h-1) (group D, n = 30) to the end of surgery.

Data collected included intraoperative and postoperative opioid consumption. Postoperative questionare including PONV, Pain intensity, I-FEED questionnaire. Prospective analysis will be performed on the prospectively collected data.

We expected to examine if intraoperative dexmedetomidine decreases the postoperative opioid consumption and associated complications, and enhances the gastrointestinal recovery and oral intake with narcotic-sparing effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfill the criteria of breast cancer under general anesthesia.

Exclusion Criteria:

* Major systemic disease, such as congestive heart failure, liver cirrhosis, end stage renal disease and malignancy.
* Patients who have the risk of difficult ventilation or intubation.
* Pregnant women.
* Coagulopathy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | postoperative 7 days
  postoperative morphine consumption by mg

SECONDARY OUTCOMES:
i-feed score | up to postoperative day 7
  recovery of eating by I-feed questionare ( score: 0-14), minimum 0 (complete recovery without eating problems), maximum 14

OTHER OUTCOMES:
changes of OCTT (orocecal transit time) by minutes | preoperative and postoperative day 1
  detect the hydrogen in exhaled gas every 15 minutes after drinking 10 gram lactulose. The time with hydrogen production more than 10 ppm is the OCTT. The changes of OCTT time between pre-operation and POD1

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to the ethical concern, we did not share our paatients' data.